CLINICAL TRIAL: NCT05441891
Title: Effect of an Equalizer-modulated Auditory Intervention on the Asymmetry of Interaural Auditory Perception in Groups of Different Emotional States
Brief Title: Effect of Modulated Auditory Stimulation on Interaural Auditory Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Francisco Germain, Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CREC/UH/2022/05
Record Dates: First submitted 2022-06-22; First posted 2022-07-01 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Asymmetric Sensorineural Hearing Loss
Keywords: hearing asymmetry; mental disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, parallel, pre-post study design
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants not received any intervention. The researchers in charge of outcome assessment and statistical analysis are blinded to the allocation of participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants assigned to the control group are cited to the Health centre, but they do not suffer any intervention. These subjects followed the same evaluation and data collection process.
- Auditory intervention filter-modulated (Active Comparator): Participants assigned to this group listened classical music modulated by an equalizer for 30 minutes, 2 sessions a day separated by at least 3 hours, for 10 days (Monday to Friday for 2 weeks).
  Interventions: Other: Auditory intervention filter-modulated group

INTERVENTIONS:
Other: Auditory intervention filter-modulated group — Intervention consisted of listening to classical music modulated by an equalizer for 30 minutes, 2 sessions a day separated by at least 3 hours, for 10 days (Monday to Friday for 2 weeks).
  The musical intervention was always performed with the same songs and in the same order using original CDs, heard through headphones (Beyerdynamic, DT 250 / 80 ohm. GMBH & Co. KG, Theresienstr. 8 D-74072 Heilbronn, Germany). The music was played with a sound system (Panasonic MASH, No. SA-PM24. Hamburg, Germany). and filtered through an equalizer called Earducator (Hollagen Designs, PÍO. Box 43 7864 Bergvliet W.Cape - South Africa) that modulates music by alternating low and high tones with an unpredictable cadence, preventing habituation. It also allows very narrow band complementary filters to attenuate (by about 40 dB) abnormally perceived frequencies (hyper-hearing peaks): filters in: 1 kHz - 1,5 kHz - 2kHz - 3 kHz - 4 kHz - 8kHz.
  Other Names: Bérard´s method
  Arms: Auditory intervention filter-modulated

SUMMARY:
This study analyzes the effect of an equalizer-modulated auditory intervention on the asymmetry of interaural auditory perception in groups with different emotional states such as well-being, anxiety, depression and mixed anxiety-depression.

DETAILED DESCRIPTION:
The present study follows a randomized, double-blind (investigator and outcome assessor), parallel and controlled design. The auditory intervention consisted of listening to classical music modulated by an equalizer for 30 minutes, 2 sessions a day separated by at least 3 hours, for 10 days (Monday to Friday for 2 weeks). Participants assigned to the control group are cited to the Health centre, but they do not received any intervention. These subjects follow the same evaluation and data collection process.

Once randomized, all participants will make a first control visit in which a pure-tone audiometry was carry out and completed the various psychiatric evaluation tests to classify into different groups: Goldberg Anxiety and Depression Scale (GADS), Hamilton Anxiety Rating Scale (HAM-A), Hamilton Depression Rating Scale (HAM-D), and Sociodemographic variables (age, gender, nationality, education, working status, noise exposure, use of ear protection, and present or past use of any analgesic, anxiolytic or antidepressant for longer than a week).

The study variables collected at 3 months were pure-tone audiometry (air conduction).

ELIGIBILITY:
Inclusion Criteria:

* Recruited from Health Centre Mejorada del Campo (Madrid, Spain)

Exclusion Criteria:

* Having significant hearing loss
* Having acute otological process
* Having psychotic disease
* Having epilepsy
* Having serious illness
* Having pregnancy
* Used to try alcohol or drugs

Ages: 31 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Change from Baseline hearing threshold at a frequency of 125 Hz in an air conduction pure tone audiometry at three months | Change from Baseline hearing threshold at 3 months
  Minimum number of decibels needed to hear a sound at a frequency of 125 Hz measured in an air conduction pure tone audiometry
Change from Baseline hearing threshold at a frequency of 250 Hz in an air conduction pure tone audiometry at three months | Change from Baseline hearing threshold at 3 months
  Minimum number of decibels needed to hear a sound at a frequency of 250 Hz measured in an air conduction pure tone audiometry
Change from Baseline hearing threshold at a frequency of 500 Hz in an air conduction pure tone audiometry at three months | Change from Baseline hearing threshold at 3 months
  Minimum number of decibels needed to hear a sound at a frequency of 500 Hz measured in an air conduction pure tone audiometry
Change from Baseline hearing threshold at a frequency of 750 Hz in an air conduction pure tone audiometry at three months | Change from Baseline hearing threshold at 3 months
  Minimum number of decibels needed to hear a sound at a frequency of 750 Hz measured in an air conduction pure tone audiometry
Change from Baseline hearing threshold at a frequency of 1000 Hz in an air conduction pure tone audiometry at three months | Change from Baseline hearing threshold at 3 months
  Minimum number of decibels needed to hear a sound at a frequency of 1000 Hz measured in an air conduction pure tone audiometry
Change from Baseline hearing threshold at a frequency of 1500 Hz in an air conduction pure tone audiometry at three months | Change from Baseline hearing threshold at 3 months
  Minimum number of decibels needed to hear a sound at a frequency of 1500 Hz measured in an air conduction pure tone audiometry
Change from Baseline hearing threshold at a frequency of 2000 Hz in an air conduction pure tone audiometry at three months | Change from Baseline hearing threshold at 3 months
  Minimum number of decibels needed to hear a sound at a frequency of 2000 Hz measured in an air conduction pure tone audiometry
Change from Baseline hearing threshold at a frequency of 3000 Hz in an air conduction pure tone audiometry at three months | Change from Baseline hearing threshold at 3 months
  Minimum number of decibels needed to hear a sound at a frequency of 3000 Hz measured in an air conduction pure tone audiometry
Change from Baseline hearing threshold at a frequency of 4000 Hz in an air conduction pure tone audiometry at three months | Change from Baseline hearing threshold at 3 months
  Minimum number of decibels needed to hear a sound at a frequency of 4000 Hz measured in an air conduction pure tone audiometry
Change from Baseline hearing threshold at a frequency of 6000 Hz in an air conduction pure tone audiometry at three months | Change from Baseline hearing threshold at 3 months
  Minimum number of decibels needed to hear a sound at a frequency of 6000 Hz measured in an air conduction pure tone audiometry
Change from Baseline hearing threshold at a frequency of 8000 Hz in an air conduction pure tone audiometry at three months | Change from Baseline hearing threshold at 3 months
  Minimum number of decibels needed to hear a sound at a frequency of 8000 Hz measured in an air conduction pure tone audiometry
Anxiety and depression level on the Goldberg scale | One month
  To discriminate between these two entities. The following cut-off points were used: a total Anxiety score > 4 detects 73% of all cases of anxiety; a total Depression score >3 detects 82% of all cases of depression
Anxiety level on the Hamilton scale | One month
  It is a clinician-administered scale on which each item is rated from 0 to 4. It yields a score in the range of 0 to 56. The following cut-off points were used: 0-5 points (No anxiety), >5 points (Anxiety).
Depression level on the Hamilton scale | One month
  Each item is rated on a three- or five-point scale, with a score from 0 to 2 or 0 to 4, respectively. It yields a total score in the range of 0 to 52. The following cut-off points were used to assess depression: No depression: 0-7; Depression: >7

SECONDARY OUTCOMES:
Relationship between the auditory threshold of the right and left ear at the frequency of 125 Hz | Three months between the first and second measure
  Ratio of the threshold of one ear to that of the other. If both have the same threshold, the result is zero.
Relationship between the auditory threshold of the right and left ear at the frequency of 250 Hz | Three months between the first and second measure
  Ratio of the threshold of one ear to that of the other. If both have the same threshold, the result is zero.
Relationship between the auditory threshold of the right and left ear at the frequency of 500 Hz | Three months between the first and second measure
  Ratio of the threshold of one ear to that of the other. If both have the same threshold, the result is zero.
Relationship between the auditory threshold of the right and left ear at the frequency of 750 Hz | Three months between the first and second measure
  Ratio of the threshold of one ear to that of the other. If both have the same threshold, the result is zero.
Relationship between the auditory threshold of the right and left ear at the frequency of 1000 Hz | Three months between the first and second measure
  Ratio of the threshold of one ear to that of the other. If both have the same threshold, the result is zero.
Relationship between the auditory threshold of the right and left ear at the frequency of 1500 Hz | Three months between the first and second measure
  Ratio of the threshold of one ear to that of the other. If both have the same threshold, the result is zero.
Relationship between the auditory threshold of the right and left ear at the frequency of 2000 Hz | Three months between the first and second measure
  Ratio of the threshold of one ear to that of the other. If both have the same threshold, the result is zero.
Relationship between the auditory threshold of the right and left ear at the frequency of 3000 Hz | Three months between the first and second measure
  Ratio of the threshold of one ear to that of the other. If both have the same threshold, the result is zero.
Relationship between the auditory threshold of the right and left ear at the frequency of 4000 Hz | Three months between the first and second measure
  Ratio of the threshold of one ear to that of the other. If both have the same threshold, the result is zero.
Relationship between the auditory threshold of the right and left ear at the frequency of 6000 Hz | Three months between the first and second measure
  Ratio of the threshold of one ear to that of the other. If both have the same threshold, the result is zero.
Relationship between the auditory threshold of the right and left ear at the frequency of 8000 Hz | Three months between the first and second measure
  Ratio of the threshold of one ear to that of the other. If both have the same threshold, the result is zero.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Estalayo-Gutierrez, MD, PhD, Principal Investigator — University of Alcalá
Locations (1):
- University of Alcalá, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frassle S, Paulus FM, Krach S, Schweinberger SR, Stephan KE, Jansen A. Mechanisms of hemispheric lateralization: Asymmetric interhemispheric recruitment in the face perception network. Neuroimage. 2016 Jan 1;124(Pt A):977-988. doi: 10.1016/j.neuroimage.2015.09.055. Epub 2015 Oct 9. PMID 26439515
- [Background] Brancucci A, Babiloni C, Rossini PM, Romani GL. Right hemisphere specialization for intensity discrimination of musical and speech sounds. Neuropsychologia. 2005;43(13):1916-23. doi: 10.1016/j.neuropsychologia.2005.03.005. Epub 2005 Mar 21. PMID 16168732